CLINICAL TRIAL: NCT06450028
Title: Lidocaine Versus Bupivacaine in Orthognathic Surgery: A Randomized Controlled Trial
Brief Title: Lidocaine Versus Bupivacaine in Orthognathic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Green, Oral and Maxillofacial Surgeon, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00047452
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Numbness; Temperature Sensation; Perception of Touch
Keywords: orthognathic surgery; lidocaine; bupivacaine; Le Fort I; bilateral sagittal split osteotomy (BSSO)
MeSH Terms: conditions — Pain, Postoperative; Hypesthesia | interventions — Bupivacaine; Epinephrine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups. Group 1 will receive 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine on the left side of their jaw and 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine on the right side of their jaw. Group 2 will receive 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine on the right side of their jaw and 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine on the left side of their jaw.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not know which anesthetic they received on each side of their jaw. The care provider, who will be administering the anesthetic intraoperatively, will know which anesthetic is being administered on each side of the participant's jaw. The outcomes assessor will not know which anesthetics was administered on each side of the participant's jaw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine Left, Lidocaine Right (Active Comparator): Group 1 will receive 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine on the left side of their jaw and 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine on the right side of their jaw. This dosage will be administered once as peripheral nerve blocks at the beginning of the participant's orthognathic procedure.
  Interventions: Drug: 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine; Drug: 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine
- Bupivacaine Right, Lidocaine Left (Active Comparator): Group 2 will receive 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine on the right side of their jaw and 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine on the left side of their jaw. This dosage will be administered once as peripheral nerve blocks at the beginning of the participant's orthognathic procedure.
  Interventions: Drug: 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine; Drug: 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine — Injection of 10 cc of 0.25% bupivacaine hydrochloride with 1:200,000 epinephrine.
  Other Names: Bupivacaine
Drug: 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine — Injection of 6.8 cc of 2% lidocaine hydrochloride with 1:100,000 epinephrine.
  Other Names: Lidocaine

SUMMARY:
In this research study, we want to learn more about the impact of two different local anesthetics (bupivacaine and lidocaine) on patient experience following orthognathic (jaw) surgery. Both anesthetics are within the standard of care for dental and orthognathic procedures, but can vary in how quickly they take action and how long they last. This study will provide us with a greater understanding of how anesthetic choice affect patient outcomes, and how we can strive to make these outcomes as favorable as possible.

DETAILED DESCRIPTION:
Aim 1: To determine if differences exist in patient-reported outcomes regarding the use of bupivacaine and lidocaine in orthognathic surgery.

Aim 2: To assess patient experiences with pain, numbness, light touch perception, temperature sensation and narcotic and pain medication consumption following administration of bupivacaine and lidocaine in orthognathic surgery.

Lidocaine (known as lignospan commercially) and bupivacaine (known as marcaine or sensorcaine commercially) are two local anesthetics used ubiquitously for procedures in the oral cavity. Lidocaine is known for its fast-acting properties, which can take effect within one to two minutes of administration. However, lidocaine also has a relatively short duration of action, typically lasting about one to two hours. On the other hand, bupivacaine is slightly slower acting (tales effect in 10-15 minutes) but has a much longer duration of action (up to eight hours). Both local anesthetics are used in orthognathic surgery (jaw surgery) and are within the standard of care for these procedures. Lidocaine and bupivacaine are both administered with epinephrine as an additive to reduce bleeding in the operative field and improve the depth and duration of anesthesia. Some patients may experience significant pain postoperatively if their local anesthetic is metabolized too quickly, while others may experience prolonged numbness and decreased sensation if their local anesthetic has too long of a duration of action.

Patients will be randomized into two equally sized groups. Group 1 will receive 0.25% bupivacaine hydrochloride and epinephrine 1:200,000 on the left side of their mandible and/or maxilla and 2% lidocaine hydrochloride with 1:100,000 epinephrine on the right side of their mandible and/or maxilla. Group 2 will receive 0.25% bupivacaine hydrochloride and epinephrine 1:200,000 on the right side of their mandible and/or maxilla and 2% lidocaine hydrochloride with 1:100,000 epinephrine on the left side of their mandible and/or maxilla. The use of bupivacaine and lidocaine are common practice in orthognathic surgery and are frequently used in conjunction with each other. Email reminders will be sent to the oral surgeon reminding them that their patients is enrolled in this study. Following that email, another email will be sent to the oral surgeon by another individual to inform them of which side they are able to administer which anesthetic. This allows the research staff member performing postoperative assessments to remain blinded.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an orthognathic procedure at Boston Children's Hospital
* Between the ages of 15 and 35 years old

Exclusion Criteria:

* Any patient undergoing any other procedures in addition to their orthognathic procedure during the same sedation period (extraction, bone graft, etc.).
* Any patient with a history of chronic pain.
* Any patient with a history of an allergic reaction to bupivacaine or lidocaine.
* Any patient with known neurologic changes to the lip or chin.
* Any patient not enrolled in an Enhanced Recovery After Surgery (ERAS) Protocol.
* Any patient known to be pregnant or with a positive pregnancy test prior to the procedure.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported pain | (1) four to six weeks prior to their orthognathic procedure, (2) approximately one hour after their orthognathic procedure, (3) approximately four hours after their orthognathic procedure, (4) one week after their orthognathic procedure.
  Pain will be measured by prompting participants to rank their pain on a scale (minimum 1, maximum 10; 1 meaning minimal pain and 10 meaning maximum pain) on each side of their mandible/maxilla. Patients will also be asked to subjectively describe their pain experiences on each side of their mandible/maxilla.

SECONDARY OUTCOMES:
Numbness | (1) four to six weeks prior to their orthognathic procedure, (2) approximately one hour after their orthognathic procedure, (3) approximately four hours after their orthognathic procedure, (4) one week after their orthognathic procedure.
  Participants will be asked to describe their feelings of numbness on a scale (minimum 1, maximum 10; 1 meaning minimal pain and 10 meaning maximum pain) on each side of their mandible/maxilla.
Light Touch and Directionality Perception | (1) four to six weeks prior to their orthognathic procedure, (2) approximately one hour after their orthognathic procedure, (3) approximately four hours after their orthognathic procedure, (4) one week after their orthognathic procedure.
  Participants will be tested regarding their perception of light touch using Von Frey hairs. Von Frey hairs are standardized plastic filaments that are numbered numerically representing the weight in grams that it takes to bend the filament. Von Frey's hairs will also be used to assess perception of directionality.
Temperature Sensation | (1) four to six weeks prior to their orthognathic procedure, (2) approximately one hour after their orthognathic procedure, (3) approximately four hours after their orthognathic procedure, (4) one week after their orthognathic procedure.
  Temperature sensation will be assessed by application of warm and cold water to mandible/maxilla using cotton tip applicators. Participants will be prompted to describe the temperature of the sensation they are experiencing.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Green, DDS, MD, Principal Investigator — Boston Children's Hospital, Department of Plastic and Oral Surgery
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers.

REFERENCES:
- See also: Lidocaine - StatPearls — https://www.ncbi.nlm.nih.gov/books/NBK539881/
- See also: Bupivacaine - StatPearls — https://www.ncbi.nlm.nih.gov/books/NBK532883/
- See also: Bupivacaine - Mayo Clinic — https://www.mayoclinic.org/drugs-supplements/bupivacaine-injection-route/description/drg-20406723
- See also: Bader JD, Bonito AJ, Shugars DA. Cardiovascular Effects of Epinephrine in Hypertensive Dental Patients: Summary. — https://www.ncbi.nlm.nih.gov/books/NBK11858/